CLINICAL TRIAL: NCT01259726
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Safety and Efficacy of VP 20621 for Prevention of Recurrence of Clostridium Difficile Infection (CDI) in Adults Previously Treated for CDI
Brief Title: Safety and Efficacy Study of VP20621 for Prevention of Recurrent Clostridium Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VP20621-200; 2010-020484-20 (EudraCT Number)
Record Dates: First submitted 2010-12-09; First posted 2010-12-14 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Clostridium Difficile Infection
Keywords: Diarrhea; Clostridium difficile; Clostridium infections; Signs and Symptoms Digestive; Bacterial Infections; Pharmacologic Actions
MeSH Terms: conditions — Clostridium Infections; Diarrhea; Signs and Symptoms, Digestive; Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- VP20621 Low Dose and Placebo (Experimental)
  Interventions: Biological: VP20621; Other: Placebo
- VP20621 High Dose and Placebo (Experimental)
  Interventions: Biological: VP20621; Other: Placebo
- VP20621 High Dose (Experimental)
  Interventions: Biological: VP20621

INTERVENTIONS:
Biological: VP20621 — VP20621 as oral liquid once daily for 7 days followed by placebo as oral liquid once daily for seven days
  Arms: VP20621 Low Dose and Placebo
Biological: VP20621 — VP20621 as oral liquid once daily for 7 days followed by placebo as oral liquid once daily for 7 days
  Arms: VP20621 High Dose and Placebo
Other: Placebo — 10 mL placebo once daily for 14 days
  Arms: Placebo; VP20621 High Dose and Placebo; VP20621 Low Dose and Placebo
Biological: VP20621 — VP20621 as oral liquid once daily for 14 days
  Arms: VP20621 High Dose

SUMMARY:
The objectives of this study are: (1) to evaluate the safety and tolerability of VP 20621 dosed orally for up to 14 days in adults previously treated for CDI; (2) to characterize the frequency and duration of stool colonization with the VP 20621 strain of C. difficile; (3) to evaluate the efficacy of VP 20621 for prevention of recurrence of CDI; and (4)to select a dose regimen of VP 20621 to be used in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, 18 years of age and over, who understand the risks and benefits of participation and have provided written informed consent for the study.
2. Subjects who are experiencing a first event or first recurrence of clostridium difficile (CDI) within the last 28 days and have been successfully treated with an antibiotic for CDI.
3. Subjects who are medically stable.
4. Subjects who are willing and able to comply with the study procedures and visit schedules outlined.
5. If female be post-menopausal, surgically sterile or agree to follow an acceptable method of birth control.

Exclusion Criteria:

1. Subjects who have had more than 2 episodes of CDI within the last 6 months.
2. Subjects who have been diagnosed with Inflammatory Bowel Disease,active Irritable Bowel Syndrome, celiac disease, active gastroparesis, toxic megacolon.
3. GI surgery within 6 weeks before the day of randomization
4. Have known immunodeficiency disorder, such as HIV Infection
5. Pregnant or breast feeding females.
6. Concurrent acute life-threatening diseases.
7. Inability to tolerate oral liquids.
8. Have an absolute neutrophil count < 1000/mm3 at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2011-06-27 (Actual); Primary Completion 2013-06-11 (Actual); Study Completion 2013-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (59):
- United States (42):
  - Modesto, California
  - Palm Desert, California
  - Sacramento, California
  - Aurora, Colorado
  - Hartford, Connecticut
  - Bay Pines, Florida
  - Jacksonville, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Maywood, Illinois
  - Anderson, Indiana
  - Lafayette, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Chevy Chase, Maryland
  - Detroit, Michigan
  - Grosse Pointe Woods, Michigan
  - Novi, Michigan
  - Royal Oak, Michigan
  - Sault Ste. Marie, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Butte, Montana
  - Omaha, Nebraska
  - Albany, New York
  - New York, New York
  - North Massapequa, New York
  - Syracuse, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Lima, Ohio
  - Toledo, Ohio
  - Lancaster, Pennsylvania
  - West Reading, Pennsylvania
  - Memphis, Tennessee
  - Houston, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Winchester, Virginia
  - Tacoma, Washington
- Belgium (4):
  - Aalst
  - Brussels
  - Leuven
  - Liège
- Canada (5):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Trois-Rivières, Quebec
- Germany (4):
  - Cologne
  - Hanover
  - Leipzig
  - Wilhelmshaven
- Spain (3):
  - Seville, Andalusia
  - Barcelona, Catalonia
  - Majadahonda, Communidad de Madrid
- Lugano, Switzerland

REFERENCES:
- [Derived] Gerding DN, Meyer T, Lee C, Cohen SH, Murthy UK, Poirier A, Van Schooneveld TC, Pardi DS, Ramos A, Barron MA, Chen H, Villano S. Administration of spores of nontoxigenic Clostridium difficile strain M3 for prevention of recurrent C. difficile infection: a randomized clinical trial. JAMA. 2015 May 5;313(17):1719-27. doi: 10.1001/jama.2015.3725. PMID 25942722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a total of 44 investigative sites [United states (US)=33, Canada=4, and Europe=7], and 3 of the 33 US sites did not enroll any participants (each had 1 screen failure).
Pre-assignment Details: Of the 213 participants formally screened to participate in this study, 168 participants were treated. Five participants were randomized but not treated and 40 participants were screen failures.
Groups:
- Placebo: Placebo matched to VP 20621 oral liquid once daily from Day 1 to 14.
- VP 20621 Low Dose and Placebo: VP 20621 oral liquid containing 10^4 purified spores of non-toxigenic Clostridium difficile-strain M3 (NTCD-M3; the dormant form of a live organism) once daily from Day 1 to 7 followed by placebo matched to VP 20621 oral liquid once daily from Day 8 to 14.
- VP 20621 High Dose and Placebo: VP 20621 oral liquid containing 10^7 purified spores of NTCD-M3 once daily from Day 1 to 7 followed by placebo matched to VP 20621 oral liquid once daily from Day 8 to 14.
- VP 20621 High Dose: VP 20621 oral liquid containing 10^7 purified spores of NTCD-M3 once daily from Day 1 to 14.
Period: Overall Study
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Started | 43 | 41 | 43 | 41
Treated | 40 | 37 | 41 | 39
Completed | 38 | 37 | 39 | 36
Not Completed | 5 | 4 | 4 | 5
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat-Safety (ITT-S) population was defined as all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose | Total
Number analyzed (Participants) | 43 | 41 | 43 | 41 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (19.19) | 58.2 (14.42) | 57.2 (18.46) | 60.6 (16.4) | 57.6 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 24 | 28 | 104
  Male | 17 | 15 | 19 | 13 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward, undesired, unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiological observations occurring in a study participant, regardless of causal relationship. TEAEs were defined as all AEs that start during the study drug treatment period (and up to 7 days after the last dose of the study drug) and were not seen at baseline, or were seen at baseline but increased in frequency and/or severity during the study drug treatment period (and up to 7 days after the last dose of study drug). SAE was any AE that results in any of the following outcomes: death, a life-threatening event, inpatient hospitalization or prolongation of an existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital anomaly/birth defect, other medically important events based upon appropriate medical judgement.
Time Frame: Baseline up to 7 days after the last dose of study drug (up to Week 3)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Number analyzed (Participants) | 43 | 41 | 43 | 41
Participants
  Participants with TEAEs | 37 | 33 | 34 | 31
  Participants with treatment-emergent SAEs | 3 | 1 | 1 | 2

2. Primary Outcome: Number of Participants With Positive Clostridium Difficile Stool Cultures Demonstrating Non-Toxigenic Clostridium Difficile-Strain M3
Time Frame: After study drug administration period (14 days) through Week 6
Population: ITT-S population.
Measure: Number; unit: Participants
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Number analyzed (Participants) | 43 | 41 | 43 | 41
Participants | 4 | 26 | 31 | 29
Statistical Analysis 1: Comparison: Placebo vs VP 20621 Low Dose and Placebo; Test type: Superiority or Other; p <= 0.0001, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 2: Comparison: Placebo vs VP 20621 High Dose and Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 3: Comparison: Placebo vs VP 20621 High Dose; Test type: Superiority or Other; p < 0.0001, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05

3. Secondary Outcome: Number of Participants With Clostridium Difficile Infection (CDI) Recurrence
Description: CDI recurrence was defined as at least 1 event characterized by ALL of the following: >=3 unformed (loose or watery) stools within 24 hours (data derived from Diarrhea case report form (CRF) page which was to be completed for any clinical event of diarrhea or loose/watery stool occurring between Day 1 and Week 6); a positive C. difficile stool assay, or pseudomembranes on endoscopy/surgery; and no other likely cause of the diarrhea in the opinion of the investigator.
Time Frame: Baseline (Day 1) up to Week 6
Population: ITT-S population.
Measure: Number; unit: Participants
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Number analyzed (Participants) | 43 | 41 | 43 | 41
Participants | 13 | 6 | 2 | 6
Statistical Analysis 1: Comparison: Placebo vs VP 20621 Low Dose and Placebo; Test type: Superiority or Other; p = 0.088, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 2: Comparison: Placebo vs VP 20621 High Dose and Placebo; Test type: Superiority or Other; p = 0.002, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 3: Comparison: Placebo vs VP 20621 High Dose; Test type: Superiority or Other; p = 0.088, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05

4. Secondary Outcome: Number of Participants With Use of Antibacterial Treatment for CDI
Description: Any antibacterial medication used after Day 1 for which the investigator selected the indication "antibacterial for C. difficile infection".
Time Frame: Baseline (Day 1) up to Week 6
Population: ITT-S population.
Measure: Number; unit: Participants
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Number analyzed (Participants) | 43 | 41 | 43 | 41
Participants | 14 | 6 | 4 | 7
Statistical Analysis 1: Comparison: Placebo vs VP 20621 Low Dose and Placebo; Test type: Superiority or Other; p = 0.054, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 2: Comparison: Placebo vs VP 20621 High Dose and Placebo; Test type: Superiority or Other; p = 0.008, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 3: Comparison: Placebo vs VP 20621 High Dose; Test type: Superiority or Other; p = 0.101, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05

5. Secondary Outcome: Number of Participants With Clinical Events of Diarrhea or Loose/Watery Stools
Description: Data were derived from all AEs starting on or after Day 1 for which a Diarrhea CRF page was completed.
Time Frame: Baseline (Day 1) up to Week 6
Population: ITT-S population.
Measure: Number; unit: Participants
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Number analyzed (Participants) | 43 | 41 | 43 | 41
Participants | 33 | 23 | 25 | 23
Statistical Analysis 1: Comparison: Placebo vs VP 20621 Low Dose and Placebo; Test type: Superiority or Other; p = 0.045, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 2: Comparison: Placebo vs VP 20621 High Dose and Placebo; Test type: Superiority or Other; p = 0.066, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05
Statistical Analysis 3: Comparison: Placebo vs VP 20621 High Dose; Test type: Superiority or Other; p = 0.045, Chi-squared — Treatment comparison with placebo using two-sided Chi-Square test at significance level p=0.05

6. Secondary Outcome: Time to First CDI Recurrence
Description: CDI recurrence was defined as at least 1 event characterized by ALL of the following: >=3 unformed (loose or watery) stools within 24 hours (data derived from Diarrhea CRF page which was to be completed for any clinical event of diarrhea or loose/watery stool occurring between Day 1 and Week 6); a positive C. difficile stool assay, or pseudomembranes on endoscopy/surgery; and no other likely cause of the diarrhea in the opinion of the investigator. Time of onset is from date of randomization to date of first CDI recurrence. Time to first CDI recurrence was assessed using Kaplan-Meier curve. Due to small number of subjects (<50%) with CDI recurrence, median time to event was not evaluable.
Time Frame: Baseline (Day 1) up to Week 6
Population: ITT-S population
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | VP 20621 Low Dose and Placebo | VP 20621 High Dose and Placebo | VP 20621 High Dose
Number analyzed (Participants) | 43 | 41 | 43 | 41
days | NA [NA to NA] — Due to small number of subjects (<50%) with CDI recurrence, median time to event was not evaluable. | NA [NA to NA] — Due to small number of subjects (<50%) with CDI recurrence, median time to event was not evaluable. | NA [NA to NA] — Due to small number of subjects (<50%) with CDI recurrence, median time to event was not evaluable. | NA [NA to NA] — Due to small number of subjects (<50%) with CDI recurrence, median time to event was not evaluable.

ADVERSE EVENTS:
Time Frame: Up to 26 Weeks
Groups:
- VP20621 Low Dose and Placebo; VP20621 High Dose and Placebo: VP20621: VP20621 as oral liquid once daily for 7 days followed by placebo as oral liquid once daily for 7 days Placebo: 10 mL placebo once daily for 14 days
Arm/Group | Placebo | VP20621 Low Dose and Placebo | VP20621 High Dose and Placebo | VP20621 High Dose
Serious Adverse Events (participants affected / at risk) | 8/43 | 5/41 | 8/43 | 6/41
Other Adverse Events (participants affected / at risk) | 37/43 | 31/41 | 34/43 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | VP20621 Low Dose and Placebo (N=41) | VP20621 High Dose and Placebo (N=43) | VP20621 High Dose (N=41)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Clostridial infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | VP20621 Low Dose and Placebo (N=41) | VP20621 High Dose and Placebo (N=43) | VP20621 High Dose (N=41)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 16 (25) | 6 (14) | 9 (11) | 9 (15)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2) | 3 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 30 (117) | 21 (69) | 27 (84) | 24 (82)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (3) | 5 (7)
Flatulence (Gastrointestinal disorders) | 7 (7) | 9 (11) | 10 (10) | 6 (9)
Nausea (Gastrointestinal disorders) | 4 (9) | 5 (7) | 4 (5) | 2 (2)
Clostridial infection (Infections and infestations) | 9 (13) | 2 (2) | 2 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 1 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (3) | 1 (1) | 1 (1) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 6 (11) | 4 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.